CLINICAL TRIAL: NCT01011855
Title: A Comparison of Thermal Responses Among Newborns to Proportional Versus Adaptive Heating Algorithms in Radiant Warmer Devices
Brief Title: Radiant Warmer Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never developed due to a change in business priority.
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Radiant Warmer Trial
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Radiant warmer bed sequence 1 (Active Comparator): Clinical care provided on three different types of cleared radiant warmer beds with temperature measurements taken for 20 hours on each of the three radiant warmer beds.
  Interventions: Device: GEHC IWS 4400 & Giraffe Warmer beds
- Radiant warmer bed sequence 2 (Active Comparator): Clinical care provided on three different types of cleared radiant warmer beds with temperature measurements taken for 20 hours on each of the three radiant warmer beds.
  Interventions: Device: GEHC IWS 4400 & Giraffe Warmer beds
- Radiant warmer bed sequence 3 (Active Comparator): Clinical care provided on three different types of cleared radiant warmer beds with temperature measurements taken for 20 hours on each of the three radiant warmer beds.
  Interventions: Device: GEHC IWS 4400 & Giraffe Warmer beds
- Radiant warmer bed sequence 4 (Active Comparator): Clinical care provided on three different types of cleared radiant warmer beds with temperature measurements taken for 20 hours on each of the three radiant warmer beds.
  Interventions: Device: GEHC IWS 4400 & Giraffe Warmer beds
- Radiant warmer bed sequence 5 (Experimental): Clinical care provided on three different types of cleared radiant warmer beds with infant temperature measurements taken for 20 hours on each of the three radiant warmer beds.
  Interventions: Device: GEHC IWS 4400 & Giraffe warmer beds
- Radiant warmer bed sequence 6 (Experimental): Clinical care provided on three different types of cleared radiant warmer beds with infant temperature measurements taken for 20 hours on each of the three radiant warmer beds.
  Interventions: Device: GEHC IWS 4400 & Giraffe Warmer beds

INTERVENTIONS:
Device: GEHC IWS 4400 & Giraffe Warmer beds — Clinical care provided first on a GEHC IWS 4400 bed with a proportional heater control algorithm, followed by care provided on a GEHC Giraffe Warmer bed with an adaptive heater control algorithm, followed by care on a GEHC Giraffe Warmer bed with a proportional heater control algorithm.
  Arms: Radiant warmer bed sequence 1
Device: GEHC IWS 4400 & Giraffe Warmer beds — Clinical care provided first on a GEHC IWS 4400 bed with a proportional heater control algorithm, followed by care provided on a GEHC Giraffe Warmer bed with a proportional heater control algorithm, followed by care on a GEHC Giraffe Warmer bed with an adaptive heater control algorithm.
  Arms: Radiant warmer bed sequence 2
Device: GEHC IWS 4400 & Giraffe Warmer beds — Clinical care is first provided on a GEHC Giraffe Warmer bed with an adaptive heater control algorithm, followed by care on a GEHC IWS 4400 bed with a proportional heater control algorithm, followed by care provided on a GEHC Giraffe Warmer bed with a proportional heater control algorithm.
  Arms: Radiant warmer bed sequence 3
Device: GEHC IWS 4400 & Giraffe Warmer beds — Clinical care is first provided on a GEHC Giraffe Warmer bed with an adaptive heater control algorithm, followed by care on a GEHC Giraffe Warmer bed with a proportional heater control algorithm, followed by care provided on a GEHC IWS 4400 bed with a proportional heater control algorithm.
  Arms: Radiant warmer bed sequence 4
Device: GEHC IWS 4400 & Giraffe warmer beds — Clinical care is first provided on a GEHC Giraffe Warmer bed with a proportional heater control algorithm, followed by care provided on a GEHC IWS 4400 bed with a proportional heater control algorithm, followed by care provided on a GEHC Giraffe Warmer bed with an adaptive heater control algorithm.
  Arms: Radiant warmer bed sequence 5
Device: GEHC IWS 4400 & Giraffe Warmer beds — Clinical care is first provided on a GEHC Giraffe Warmer bed with a proportional heater control algorithm, followed by care provided on a GEHC Giraffe Warmer bed with an adaptive heater control algorithm, followed by care provided on a GEHC IWS 4400 bed with a proportional heater control algorithm.
  Arms: Radiant warmer bed sequence 6

SUMMARY:
The purpose of this study is to compare three radiant warmer beds that contain different computer heating software and different bed styles. Radiant warmers are used in many neonatal intensive care units (NICU) to provide heat to infants to help regulate an infant's temperature. It is common for babies to require care on an open bed that provides heat to the baby according to the baby's needs and at the same time allows easy access to the baby for care and necessary procedures. There are different styles of beds, each with unique computer software that can guide how a bed's heater output is automatically adjusted according to a baby's temperature needs. It is unknown which style of bed or method of heating might be best. This study seeks to evaluate infant responses to three different types of radiant warmer beds.

DETAILED DESCRIPTION:
Study was withdrawn

ELIGIBILITY:
Inclusion Criteria:

* Any baby > 32 weeks gestation and > 1500 grams that requires initial care on a radiant warmer during confinement in the neonatal intensive care unit.

Exclusion Criteria:

* Any baby who has a skin condition that may prevent or compromise thermistor placement and interfere with accurate temperature readings from thermistors or IR camera.
* Any baby who is deemed too sick to tolerate movement from one radiant warmer to another by the attending physician.
* Any baby who has a medical condition or anomaly that contraindicates axillary or abdominal temperature measurements

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Abdominal skin surface temperatures and axillary temperatures under 3 radiant warmer conditions as measured by skin thermistors and infrared thermography (IRT). | There is a 4-hour baseline/washout period, followed by a 20-hour data collection cycle that will be repeated for all three-treatment conditions. Samples from the bed and telethermometer will be collected electronically every 60 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Sturtz, MD, Principal Investigator — Christiana Care